CLINICAL TRIAL: NCT04595786
Title: A Randomized, Parallel-group, Placebo Control, Non-inferiority Trial to Investigate the Safety of Intravenous Tranexamic Acid in Patients Undergoing Supratentorial Meningiomas Resection
Brief Title: The Safety of Intravenous Tranexamic Acid in Patients Undergoing Supratentorial Meningiomas Resection
Acronym: STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ChiECRCT20200224
Record Dates: First submitted 2020-10-09; First posted 2020-10-22 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Seizures; Meningioma
Keywords: meningioma; blood management
MeSH Terms: conditions — Seizures; Meningioma | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXA group (Active Comparator): The TXA group will receives Tranexamic acid intraoperative.
  Interventions: Drug: Tranexamic acid
- Placebo group (Placebo Comparator): The TXA group will receives 0.9% saline intraoperative.
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Tranexamic acid — 20mg/kg TXA was prepared in a 50ml syringe for intravenous pump
  Arms: TXA group
Drug: 0.9% saline — 0.9% saline was prepared in a 50ml syringe for intravenous pump
  Arms: Placebo group

SUMMARY:
Growing evidence of Tranexamic Acid (TXA) being used to reduce blood loss and blood transfusions in various guidelines. However, the adverse effects of TXA especially seizure has always been a problem of concern, especially in neurosurgery. Therefore, this study aims to provide a scientific evidence for the safety of TXA in supratentorial meningiomas resection patients.

ELIGIBILITY:
Inclusion Criteria:

* 1) age 18-80 years
* 2) American Society of Anesthesiologist (ASA) classification score I~III

Exclusion Criteria:

* 1) allergic to tranexamic acid
* 2) preoperative seizures
* 3) history of thrombotic disease
* 4) chronic kidney disease
* 5) breastfeeding or pregnancy
* 6) refuse to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Early postoperative seizures within 7 days | Within 7 days after surgery
  Postoperative seizures were defined as a transient occurrence of involuntary movements, abnormal sensory phenomena, or an altered mental status that could not otherwise be explained.

SECONDARY OUTCOMES:
The incidence of non-epileptic complications | Within 7 days after the intervention
  Including intracranial hematoma, deep vein thrombosis, pulmonary embolism, cerebral venous sinus thrombosis, stroke, myocardial infarction, acute kidney infarction, anaemia, and infection.
Estimated intraoperative blood loss | During surgery
  Estimated intraoperative blood loss = collected blood volume in the suction canister (ml) - volume of flushing (ml) + volume from gauze tampon (ml).
The changes in haemoglobin concentrations | During surgery
  The changes in haemoglobin concentrations between baseline and end of surgery.
The intraoperative blood transfusion volume and rate | During surgery
  The intraoperative blood transfusion volume and rate.
The intraoperative cell saver volume and rate | During surgery
  The intraoperative cell saver volume and rate.

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, M.D., Ph.D, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual, de-identified participant data will be shared two years after the publication of primary outcome data, by request from any qualified investigator following approval of a protocol, statistical analysis plan, and receipt of a signed data access agreement via the research office and the Beijing Tiantan Hospital Ethics Committees for the project and data release.
Supporting Information: Study Protocol, SAP
Time Frame: Two years after the primary outcome data is published.

REFERENCES:
- [Derived] Li S, Liu M, Yang J, Yan X, Wu Y, Zhang L, Zeng M, Zhou D, Peng Y, Sessler DI. Intravenous tranexamic acid for intracerebral meningioma resections: A randomized, parallel-group, non-inferiority trial. J Clin Anesth. 2024 Feb;92:111285. doi: 10.1016/j.jclinane.2023.111285. Epub 2023 Oct 17. PMID 37857168
- [Derived] Li S, Yan X, Li R, Zhang X, Ma T, Zeng M, Dong J, Wang J, Liu X, Peng Y. Safety of intravenous tranexamic acid in patients undergoing supratentorial meningiomas resection: protocol for a randomised, parallel-group, placebo control, non-inferiority trial. BMJ Open. 2022 Feb 2;12(2):e052095. doi: 10.1136/bmjopen-2021-052095. PMID 35110315